CLINICAL TRIAL: NCT00914433
Title: A Phase 1,Randomized, Double--blind, Placebo-controlled Study Assessing the Safety and Tolerability, the Pharmacodynamics and Pharmacokinetics of Single-ascending and Repeated Doses of Inhaled TPI 1100 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Inhaled TPI 1100 in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug development suspended
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TPI 1100-101
Record Dates: First submitted 2009-06-02; First posted 2009-06-05 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TPI 1100 (Experimental): Drug to be given by inhalation.
  Interventions: Drug: TPI 1100

INTERVENTIONS:
Drug: TPI 1100 — 1 dose only increasing dose

SUMMARY:
This study will look at the safety and tolerability of TPI 1100 in healthy volunteers and look at pharmacodynamic (PD) effect on mRNA expression of PDE 4B/D & 7A in blood and in sputum.

DETAILED DESCRIPTION:
Study was not initiated and terminated before start-up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female volunteers aged 18 to 55 years inclusive
* Screening/baseline FEV1 greater than 90% predicted,
* Body mass index (BMI) of 19 to 28 inclusive,
* Clinical laboratory values and/or vital signs within normal reference ranges or not considered clinically significant by the Investigator

Exclusion Criteria:

* Airways or systemic conditions that might affect respiratory function, including but not limited to clinically significant cardiac problems,
* Breast-feeding or pregnancy,
* Positive tests for smoking tobacco, alcohol, hepatitis B-surface antigen, hepatitis C antibody, and HIV at screening,
* History of serious adverse reaction to any drugs,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Airway-specific and general safety and tolerability. | 24 hours post-dose and on Day 4

SECONDARY OUTCOMES:
Effect on mRNA | 24 hrs post-dose and on Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Pageau, Study Director — Topigen Pharmaceuticals Inc.